CLINICAL TRIAL: NCT04901689
Title: A Phase 3, Randomized, Double Blind, Placebo Controlled Trial to Evaluate the Efficacy and Safety of Leronlimab in Combination With Standard of Care for Patients With Coronavirus Disease 2019 (COVID-19) With Need for Mechanical Ventilation or Extracorporeal Membrane Oxygenation
Brief Title: Leronlimab in Patients With Coronavirus Disease 2019 (COVID-19) With Need for Mechanical Ventilation or Extracorporeal Membrane Oxygenation
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Pending DSMB evaluation
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: CytoDyn, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARO_21_018_002
Record Dates: First submitted 2021-05-24; First posted 2021-05-25 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2021-05

CONDITIONS: COVID-19 Pneumonia
Keywords: COVID-19; Pneumonia; Leronlimab
MeSH Terms: conditions — COVID-19; Pneumonia | interventions — leronlimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Leronlimab (700 mg) (Experimental): Leronlimab 700 mg intravenously once a week (up to 4 doses) until hospital discharge
  Interventions: Drug: Leronlimab
- Placebo (Placebo Comparator): Placebo intravenously once a week (up to 4 doses) until hospital discharge
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Leronlimab — Leronlimab 700 mg
  Arms: Leronlimab (700 mg)
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Leronlimab (PRO 140) is a humanized IgG4,k monoclonal antibody (mAb) that recognizes the C-C chemokine receptor type 5 (CCR5). Disruption of the C-C chemokine ligand 5 (CCL5)-CCR5 axis via leronlimab-mediated CCR5 blockade might prevent pulmonary trafficking of pro-inflammatory leukocytes and dampen pathogenic immune activation in coronavirus disease 2019 (COVID-19).

The purpose of the study is to assess the safety and efficacy of leronlimab plus standard of care in critically ill patients hospitalized with COVID-19 pneumonia who are requiring mechanical ventilation or extracorporeal oxigenation (ECMO).

DETAILED DESCRIPTION:
Leronlimab (PRO 140) is a humanized IgG4,k monoclonal antibody (mAb) that recognizes the C-C chemokine receptor type 5 (CCR5). CCR5 is expressed predominantly on T cells but also found on macrophages, dendritic cells, and eosinophils to mediate chemotaxis in response to its cognate ligands that include CCL5 (RANTES), CCL3 (MIP-1α), and CCL4 (MIP-1β). These ligands are integral in the recruitment of these immune cells to inflammatory sites. The immunopathogenesis of COVID-19 likely involves the excessive influx of immune cells into the lung. Disruption of the CCL5-CCR5 axis via leronlimab-mediated CCR5 blockade might prevent pulmonary trafficking of pro-inflammatory leukocytes and dampen pathogenic immune activation in COVID-19.

The purpose of the study is to assess the safety and efficacy of leronlimab plus standard of care in critically ill patients hospitalized with COVID-19 pneumonia who are requiring mechanical ventilation or extracorporeal oxigenation (ECMO).

This is a Phase 3, 2-arm, randomized, double blind, placebo controlled, multicenter study to evaluate the safety and efficacy of leronlimab (PRO 140) as an add on therapy to the institutional standard of care (SoC) for the management of critically ill patients with COVID-19 pneumonia.

Patients will be randomized in a 1:1 ratio to receive up to four doses of 700 mg leronlimab (PRO 140) or placebo. Leronlimab or placebo will be administered by 30-minute intravenous (IV) infusion weekly over a 4-week treatment period. No treatments will be administered post-discharge.

The participant will be evaluated on each study day while hospitalized up until and including Day 28. The daily visits will capture clinical status - ordinal scale and the occurrence of adverse events. A complete follow-up assessment will be performed at Days 7, 14, 21, 28, 42 and 60 for those who are hospitalized at these specific timepoints. Follow-up visits can be conducted as telephone or video contact visits, if subject is discharged from the hospital prior to the complete follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Male or females aged ≥ 18 years
2. Critically ill patients with COVID-19 (defined as Ordinal Scale score of 7): Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO) for less than 72 hours.
3. Evidence of pneumonia (pulmonary infiltrates) at chest radiography or computed tomography compatible with COVID-19.
4. Laboratory-confirmed novel coronavirus (SARS-CoV-2) infection as determined by polymerase chain reaction (PCR).
5. Subject (or legally authorized representative) provides written or oral informed consent prior to initiation of any study procedures.
6. Women of childbearing potential and their partner must agree to use at least one highly effective method of contraception (e.g., hormonal contraceptives [implants, injectables, combination oral contraceptives, transdermal patches, or contraceptive rings], intrauterine devices, bilateral tubal occlusion, or sexual abstinence) for the duration of the study.

Exclusion Criteria:

1. Subjects who had been on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO) for >72 hours prior to the screening.
2. Subjects who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to leronlimab (PRO 140) are not eligible.
3. Inability to provide informed consent (from subject or legally authorized representative) or to comply with test requirements.
4. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk associated with study participation or, in the investigator's judgment, make the participant inappropriate for the study.
5. Pregnancy or breast feeding.
6. Subject participating in another study with for an investigational treatment.
7. Suspected or known active systemic bacterial, fungal, or viral infections (with the exception of COVID-19), that may increase the risk for the study participant based on investigator judgement.
8. Participants who are immunocompromised, with known immunodeficiencies, or taking potent immunosuppressive agents (e.g., azathioprine, cyclosporine).
9. Patients with estimated discharge or transfer for other hospital in the first 72 hours of study inclusion.
10. Patients with low probability of survival in the first 48 hours of study inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2021-10-23 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Cumulative proportion of clinical recovery | 28 days
  Patients will be considered to have recovered if they attain categories 1, 2, or 3 on the eight-category ordinal scale within 28 days, as follows:
  1. Not hospitalized, no limitations on activities
  2. Not hospitalized, limitation on activities and/or requiring home oxygen
  3. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care
  4. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise)
  5. Hospitalized, requiring supplemental oxygen
  6. Hospitalized, on non-invasive ventilation or high flow oxygen devices
  7. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO)
  8. Death

SECONDARY OUTCOMES:
Proportion of patients clinically recovered | At days 14, 28, 42, and 60
  Ordinal Scale of 1, 2 or 3
All-cause mortality | At days 14, 28, 42, and 60
  All-cause mortality
Proportion of patients discharged alive | At days 14, 28, 42, and 60
  Ordinal Scale 1 or 2
Clinical Status | Days 14, 28, 42, and 60
  Ordinal Scale
Duration of invasive mechanical ventilation or ECMO | 28 days
  Days
Length of hospital stay | 28 days
  Days
Length of ICU stay | 28 days
  Days

CONTACTS AND LOCATIONS:
Locations (23):
- Brazil (23):
  - Hospital Dr Jayme dos Santos Neves, Laranjeiras, Espírito Santo
  - Clinica São Roque, Ipiaú, Estado de Bahia
  - Santa Casa de Misericórdia da Bahia - Hospital Santa Izabel, Salvador, Estado de Bahia
  - Hospital do Coração do Brasil, Brasília, Federal District
  - Santa Casa de Misericórdia de Passos, Passos, Minas Gerais
  - Hospital 9 de Julho, São Paulo, Please Select
  - Hospital São Lucas Copacabana, Rio de Janeiro, Rio de Janeiro
  - Instituto Atena de Pesquisa Clínica, Natal, Rio Grande do Norte
  - Hospital São Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Hospital Mãe de Deus, Porto Alegre, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericórdia Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisa Clínica do Coração, Aracaju, Sergipe
  - Fundação PIO XII, Barretos, São Paulo
  - Irmandade do Sr. Bom Jesus dos Passos da Santa Casa de Misericórdia de Bragança Paulista, Bragança Paulista, São Paulo
  - Instituto de Pesquisa Clínica de Campinas, Campinas, São Paulo
  - Hospital Santa Ignes, Indaiatuba, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo
  - BP Mirante, São Paulo, São Paulo
  - Hospital Alemão Oswaldo Cruz, São Paulo, São Paulo
  - Hospital Beneficência Portuguesa, São Paulo, São Paulo
  - Santa Casa de Votuporanga, Votuporanga, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo
  - Hospital M'Boi Mirim, São Paulo

IPD SHARING:
Plan to Share IPD: No